CLINICAL TRIAL: NCT03126942
Title: Single-implant Overdentures Retained by the Novaloc Attachment System: Study Protocol for a Mixed Methods Randomized Cross-over Trial
Brief Title: Single-implant Overdentures Retained by the Novaloc Attachment System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University (Other)
Collaborators: ITI International Team for Implantology, Switzerland (Other); Institut Straumann AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: A03-M07-17A; 1185_2016 (Other Grant/Funding Number: ITI - International Team for Implantology)
Record Dates: First submitted 2017-04-13; First posted 2017-04-25 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Edentulous Mouth; Edentulous Jaw
Keywords: Aged patients; Cost Estimates; Complete Denture; Dental Economics; Dental Implants; Dental Prosthesis, Implant-Supported; Denture Retention; Minimally Invasive Surgical Procedures; Oral Health-Related Quality of Life; Overdenture; Patient Acceptance of Health Care; Quality of Healthcare; Quality of Life; Patient Satisfaction; Single implant overdenture
MeSH Terms: conditions — Mouth, Edentulous; Jaw, Edentulous; Patient Acceptance of Health Care; Patient Satisfaction

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Novaloc, then Locator (Experimental): Participants will receive the Novaloc attachment on a single implant inserted in the mandibular midline. This attachment will be used for 3 months and then changed by the Locator attachment. The second attachment will be used for another 3-month period. Participants will keep preferred attachment for further 12 months
  Interventions: Device: Novaloc; Device: Locator
- Locator, then Novaloc (Active Comparator): Participants will receive the Locator attachment on a single implant inserted in the mandibular midline. This attachment will be used for 3 months and then changed by the Novaloc attachment. The second attachment will be used for another 3-month period. Participants will keep preferred attachment for further 12 months
  Interventions: Device: Novaloc; Device: Locator

INTERVENTIONS:
Device: Novaloc — Attachment composed by a polyetheretherketone (PEEK) capsule and carbon-coated abutment. The yellow (medium) retentive component will be used
Device: Locator — Traditional cylindrical attachment (Locator system) with pink (medium) retentive components

SUMMARY:
The objective of this explanatory mixed methods study is to compare a novel attachment system (Novaloc) to a traditional alternative (Locator) for single implants in the mandible of edentate elders. The investigators will carry out a randomized cross-over clinical trial comparing Novaloc attachments to Locators for single-implant mandibular overdentures in edentate elders. Participants will be followed for three months with each attachment type; patient-based, clinical and economic outcomes will be gathered. A sample of 26 participants is estimated to be required to detect clinically relevant differences in terms of the primary outcome (patient ratings of general satisfaction). Participants will choose which attachment they wish to keep, then be interviewed about their experiences and preferences with a single implant prosthesis and with the 2 attachments. Data from the quantitative and qualitative assessments will be integrated through a mixed-methods explanatory strategy. A last quantitative assessment will take place after 12 months with preferred attachment; this latter assessment will enable the observation of attachments' long-term wear and maintenance events.

ELIGIBILITY:
Inclusion Criteria:

* Not have had a tooth extraction within the past six months
* Request implant stabilization of a mandibular conventional complete denture
* Have clinically acceptable maxillary and mandibular complete dentures
* Have adequate bone in the anterior mandible for the placement of a single 3.3 mm wide implant in the midline
* Be able to maintain adequate oral hygiene and clean dentures;
* Present no systemic conditions for which minor oral surgery would be counter-indicated
* Have an adequate understanding of written and spoken English or French;
* Be capable of giving written informed consent

Exclusion Criteria:

* Severe/serious illness that requires frequent hospitalization
* Impaired cognitive function
* Unable to return for evaluations/study recalls
* Have a history of radiation therapy to the orofacial region
* Have specific conditions that may jeopardize the treatment, such as alcoholism or smoking (>10 cigarettes/day)
* Have acute or chronic symptoms of parafunctional or temporomandibular disorders
* Previous dental implant treatment

Following radiographic exam, investigators will exclude volunteers with bony pathologic lesions, less than 11 mm of minimum vertical mandibular bone height in the midline or width for planned implants, evident endosseous vascular structures or mandibular ridges with remaining alveolar sockets

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2021-03-08 (Actual)

PRIMARY OUTCOMES:
Denture satisfaction | 18 months
  To be assessed by specific questionnaires

SECONDARY OUTCOMES:
Oral health-related quality of life | 18 months
  To be assessed by the OHIP-EDENT (Oral Health Impact Profile, shortened version for edentulous subjects) questionnaire
Overdenture rotation | 18 months
  Two questions regarding perceived rotation, as done by Kimoto et al. (Clin Oral Implants Res 2009;20:838-43)
Success/survival rate | 18 months
  Success/survival rate of prostheses and implants (yes/no)
Plaque Index | 18 months
  Presence of plaque according to Silness & Loe (Acta Odont Scand 1963;21:533-51) (ordinal scale ranging from 0 to 3)
Presence of calculus | 18 months
  Presence of calculus according to Ramfjord (J Periodontol 1967;38:602-10) (ordinal scale ranging from 0 to 3)
Peri-implant probing depth | 18 months
  Depth of peri-implant pockets (in mm)
Bleeding on probing | 18 months
  Bleeding on probing around implant (yes/no)
Mucosal inflammation | 18 months
  Signs of swelling or inflammation of the peri-implant-mucosa (yes/no, plus categorical evaluation - type of pathological change)
Treatment costs | 18 months
  Specific forms quantifying costs involved with cost of labor, materials, radiographs, medications, patient's time and transportation expenses

OTHER OUTCOMES:
Qualitative assessment | 6 months
  Qualitative assessment (descriptive approach based on transcribed interviews) regarding: a) patients' reasons for choosing one attachment system; b) their perceptions of the advantages and disadvantages of each attachment; and c) their experience of living with a single implant retention for their mandibular overdenture

CONTACTS AND LOCATIONS:
Overall Officials: Raphael F de Souza, Principal Investigator — McGill University, Faculty of Dentistry
Locations (1):
- McGill University, Faculty of Dentistry, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] de Souza RF, Jabbar AA, Jafarpour D, Bedos C, Esfandiari S, Makhoul NM, Dagdeviren D, Abi Nader S, Feine JS. Single-Implant Overdentures Retained by a Novel Attachment: A Mixed Methods Crossover Randomized Clinical Trial. JDR Clin Trans Res. 2024 Jan;9(1):27-41. doi: 10.1177/23800844221124083. Epub 2022 Sep 20. PMID 36127832
- [Derived] de Souza RF, Bedos C, Esfandiari S, Makhoul NM, Dagdeviren D, Abi Nader S, Jabbar AA, Feine JS. Single-implant overdentures retained by the Novaloc attachment system: study protocol for a mixed-methods randomized cross-over trial. Trials. 2018 Apr 23;19(1):243. doi: 10.1186/s13063-018-2606-7. PMID 29685161